CLINICAL TRIAL: NCT04358939
Title: Evaluation of Prone Position in Conscious Patients on Nasal High-flow Oxygen Therapy for COVID-19 Disease Induced Acute Respiratory Distress Syndrome
Brief Title: Prone Position in Patients on High-flow Nasal Oxygen Therapy for COVID-19 (HIGH-PRONE-COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIGH-PRONE-COVID-19; 2020-A01121-38 (Other: IdRCB); DR200125 (Other: University Hospital, Tours)
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19
Keywords: Acute Respiratory Distress Syndrome; COVID-19; SARS-CoV-2; Nasal High-Flow; Prone position
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone decubitus group (Experimental): Prone positioning of patients on nasal high-flow oxygen therapy with usual care
  Interventions: Other: Prone decubitus
- Control group (No Intervention): Patients on nasal high-flow oxygen therapy with usual care and positioned in supine

INTERVENTIONS:
Other: Prone decubitus — According to the tolerance, the objective is to spend as much time as possible, up to 16 hours and beyond in prone position every 24 hours. At least two sessions of at least 30 minutes each must be performed daily.
  Arms: Prone decubitus group

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) induces high mortality, particularly in the context of COVID-19 disease. Preliminary data from patients with ARDS related to COVID-19 disease appear to show significant effectiveness of prone positioning in intubated patients in terms of oxygenation as well as nasal high flow therapy before intubation. It should be noted that in Jiangsu province, secondarily affected, nasal high flow combined with the prone position was successfully integrated into care protocols.

The investigators hypothesize that the combined application of nasal high flow and prone positioning can significantly improve the outcome of patients suffering from COVID-19 pneumonia by reducing the need for tracheal intubation and associated therapeutics such as sedation and paralysis, resulting in both individual and collective benefits in terms of use of scarce critical care resources.

Investigators hypothesize that the combined application of nasal high-flow and prone positioning can significantly improve the outcome of patients suffering from COVID-19 pneumonia by reducing the need for intubation and associated therapeutics such as sedation and paralysis, resulting in both individual and collective benefits in terms of use of scarce critical care resources.

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) induces high mortality, particularly in the context of COVID-19 disease. In patients with ARDS who are mechanically ventilated invasively through a tracheal tube and with a PaO2/FiO2 ratio (arterial oxygen partial pressure to inspired oxygen fraction ratio) of less than 150 mmHg, prone positioning significantly reduced mortality. Furthermore, nasal high flow, a non-invasive respiratory support and oxygenation technique, reduced the need for tracheal intubation and reduced mortality among the most severe patients (PaO2/FiO2 ratio less than 200 mmHg) suffering from acute hypoxemic respiratory failure. Prone positioning of ARDS patients treated with nasal high-flow was evaluated in 20 patients with predominantly viral pneumonia. The prone positioning was found to be feasible and associated with an increased PaO2/FiO2 ratio. Preliminary data from patients with ARDS related to COVID-19 disease appear to show a significant effect of prone positioning in intubated patients in terms of oxygenation improvement as well as nasal high-high flow appears effective in non-intubated patients. For instance, nearly half intensive care unit patients described in the princeps cohort in Wuhan City, Hubei Province, China, had received nasal high-flow. It should be noted that in Jiangsu province, secondarily affected, nasal high-flow combined with prone positioning was successfully integrated into care protocols.

Investigators hypothesize that the combined application of nasal high-flow and prone positioning can significantly improve the outcome of patients suffering from COVID-19 pneumonia by reducing the need for intubation and associated therapeutics such as sedation and paralysis, resulting in both individual and collective benefits in terms of use of scarce critical care resources.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* with COVID-19 pneumonia according to the diagnostic criteria in effect at the time of inclusion or very highly suspected.
* Patient treated with nasal high-flow
* Mild, moderate or severe ARDS: bilateral radiological opacities not fully explained by effusions, atelectasis or nodules; acute hypoxemia with worsening within the previous 7 days, not fully explained by left ventricular failure; PaO2/FiO2 ratio < 300 mmHg (or equivalent SpO2/FiO2).
* Covered by or having the rights to French social security
* Informed Consent

Exclusion Criteria:

Pregnant or breastfeeding woman

* Indication for immediate tracheal intubation
* Progressive significant acute circulatory insufficiency
* Impaired alertness, confusion, restlessness
* Body mass index > 40 kg/m2
* Thoracic trauma or other contraindication to prone position
* Pneumothorax with single anterior thoracic drain and persistent bubbling
* Vulnerable person: safeguard of justice, guardianship or authorship known at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Therapeutic failure within 14 days of randomization | From randomization to day 14
  Therapeutic failure is defined by death or intubation or use of non-invasive ventilation at two pressure levels.

SECONDARY OUTCOMES:
Therapeutic failure within 28 days of randomization | From randomization to day 28
  Therapeutic failure is defined by death or intubation or use of non-invasive ventilation at two pressure levels.
Timeframe of intubation or death | From randomization to day 28
Timeframe of therapeutic escalation (in case of non-invasive ventilation at two pressure levels) | From randomization to day 28
Evolution of oxygenation (PaO2/FiO2 ratio or SpO2/FiO2 surrogate) over the 14 days following randomization | From randomization to day 14
Evolution of the SpO2/FiO2 ratio during the first prone session | From randomization to day 1
Evolution of the ROX index during the first prone session | From randomization to day 1
  ROX index is the ratio of pulse oximetry (SpO2)/fraction of inspired oxygen (FiO2) to respiratory rate.
Evolution of the World Health Organization disease severity score of COVID | From randomization to day 28
  Score reaches from 1 to 7, 7 indicates worse outcome
Patient comfort before, during and after the first prone position session | From randomization to day 1
  Comfort evaluted by the patient through a visual analogical scale
Occurrence of skin lesions on the anterior surface of the body | From randomization to day 28
Displacement of invasive devices during reversals | From randomization to day 28
  Invasive devices include : central and peripheric vascular catheters, tracheal tube, urinary catheter, chest tubes.
Days of nasal High-Flow therapy use in the general population, in non-intubated patients and in intubated patients | From randomization to day 28
Days spent in the intensive care unit and in the hospital | From randomization to day 28
Mortality in the intensive care unit and in the hospital | From randomization to day 28
Ventilator-free-days within 28 days of randomization | From randomization to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Yonatan PEREZ, MD, Study Director — No affiliation
Locations (24):
- France (24):
  - Intensive Care Unit, University Hospital, Aix, Aix-en-Provence
  - Medical Intensive Care Unit, University Hospital, Amiens, Amiens
  - Intensive Care Unit, Hospital, Argenteuil, Argenteuil
  - Medical Intensive Care Unit, Hospital, Béthune, Béthune
  - Intensive Care Unit, Hospital,, Blois
  - Medical Intensive Care Unit, University Hospital, Brest, Brest
  - Medical Intensive Care Unit, University Hospital, Caen, Caen
  - Intensive Care Unit, Louis Mourier-APHP, Colombes
  - Intensive Care Unit, Hospital, Dax, Dax
  - Medical Intensive Care Unit, University Hospital, Dijon, Dijon
  - Medical Intensive Care Unit, University Hospital, Grenoble, Grenoble
  - Intensive Care Unit, Hospital, La Roche-sur-Yon, La Roche-sur-Yon
  - Intensive Care Unit, Hospital, Le Mans, Le Mans
  - Intensive Care Unit, University Hospital, Lille, Lille
  - Medical Intensive Care Unit, University Hospital, Nantes, Nantes
  - Medical Intensive Care Unit, University Hospital, Nice, Nice
  - Medical Intensive Care Unit, Hospital, Orléans, Orléans
  - Medical Intensive Care Unit, Tenon-APHP, Paris
  - Medical Intensive Care Unit, University Hospital, Poitiers, Poitiers
  - Medical Intensive Care Unit, University Hospital, Tours, Tours
  - Surgical Intensive Care Unit, University Hospital, Tours, Tours
  - Intensive Care Unit, Hospital, Valence, Valence
  - Medical Intensive Care Unit, University Hospital, Nancy, Vandœuvre-lès-Nancy
  - Intensive Care Unit, Hospital, Vannes, Vannes

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification can be obtained by contacting the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available immediately following publication and ending in 5 years.
Access Criteria: Contact with the corresponding author.

REFERENCES:
- [Result] Ehrmann S, Li J, Ibarra-Estrada M, Perez Y, Pavlov I, McNicholas B, Roca O, Mirza S, Vines D, Garcia-Salcido R, Aguirre-Avalos G, Trump MW, Nay MA, Dellamonica J, Nseir S, Mogri I, Cosgrave D, Jayaraman D, Masclans JR, Laffey JG, Tavernier E; Awake Prone Positioning Meta-Trial Group. Awake prone positioning for COVID-19 acute hypoxaemic respiratory failure: a randomised, controlled, multinational, open-label meta-trial. Lancet Respir Med. 2021 Dec;9(12):1387-1395. doi: 10.1016/S2213-2600(21)00356-8. Epub 2021 Aug 20. PMID 34425070
- [Result] Ibarra-Estrada M, Li J, Laffey JG, Pavlov I, Roca O, Perez Y, McNicholas B, Vines D, Tavernier E, Ehrmann S. Prone positioning might reduce the need for intubation in people with severe COVID-19 - Authors' reply. Lancet Respir Med. 2021 Dec;9(12):e111. doi: 10.1016/S2213-2600(21)00449-5. No abstract available. PMID 34861160
- [Result] Tavernier E, McNicholas B, Pavlov I, Roca O, Perez Y, Laffey J, Mirza S, Cosgrave D, Vines D, Frat JP, Ehrmann S, Li J. Awake prone positioning of hypoxaemic patients with COVID-19: protocol for a randomised controlled open-label superiority meta-trial. BMJ Open. 2020 Nov 11;10(11):e041520. doi: 10.1136/bmjopen-2020-041520. PMID 33177145